CLINICAL TRIAL: NCT01640223
Title: SEMI-CLOSED LOOP "FOR THE CONTROL OF BLOOD GLUCOSE IN DIABETIC SUBJECTS DIABELOOP First CLINICAL PROJECT: Under Project 3 (UP3), CREATING A DATABASE
Brief Title: Creation of a Patient Database for Silicon Patient Simulation, Glucose Sensor Variability and Pharmacokinetic Study of Debiotech Jewelpump
Acronym: DiabeloopWP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A00726-35
Record Dates: First submitted 2012-07-05; First posted 2012-07-13 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-3 sensor (Experimental): patients will be equiped with 2 Dexcom sensors 3 days before hospitalization
  Interventions: Device: Dexcom7
- D-1 sensor (Experimental): patients will be equiped with 2 Dexcom sensors one day before hospitalization
  Interventions: Device: Dexcom7

INTERVENTIONS:
Device: Dexcom7 — patients will wear 2 Dexcom sensors 3 days before hospitalization.
  Arms: D-3 sensor
Device: Dexcom7 — patients will wear 2 Dexcom sensor one day before hospitalization
  Arms: D-1 sensor

SUMMARY:
The aim this study is the acquisition and management of a data base for the development of the glycaemic regulation algorithms. This database will integrate the measures of blood glucose and the glycaemia level of the Dexcom sensor on a regular time, the injections of insulin delivered by Debiotech JewelPUMP and the level of insulin in the blood. This database will also contain the bolus of insulin injected at meals and the content of meals, the reduction insulin level during physical activity and the quantification of this physical activity. A study will also be conducted to compare the pharmacokinetics of a bolus of insulin identical with the JewelPUMP either the usual pump of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes type 1 Treaty by external insulin pump
* Duration of diabetes than 2 years or c indosable peptide
* Practicing insulin functional (IF) or food plan sets
* Patient having a HbA1c < 10%
* Patient age over 18 years
* Patient having signed the form of collection of free consent and informed
* Patient affiliated with the social security

Exclusion Criteria:

* Patients with diabetes type 2
* Patient pregnant or likely to be
* All serious pathologies that can interfere with the study (in particular kidney or heart failure)
* Psychiatric pathologies incompatible with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Percentage of data collected | Blood glucose and insuline will be collected during the hospital stay of patient (in average 25 hours)
  The aim of the study is data collection of patient blood glucose and insulin in patients treated with continuous subcutaneous infusion insulin pump with a patchpump (JewelPUMPTM Debiotech) and equipped with two glucose sensors for the development of the control algorithm glucose.
  Blood sample are done every hour (achievement of glucose and insulin assays) ans every 15 minutes during 2 hours after meals.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHARPENTIER, MD, Study Chair — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète; Bruno GUERCI, MD PHD, Principal Investigator — Central Hospital, Nancy, France
Locations (7):
- France (7):
  - Chu Montpellier, Montpellier, Montpellier
  - CHU Toulouse, Toulouse, Toulouse
  - CHU Jean Minjoz, Besançon
  - CHU de Caen, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - University Hospital Grenoble, Grenoble
  - CHU de Nancy, Nancy